CLINICAL TRIAL: NCT01089335
Title: Sentinel Node Investigation in Patients With Highly Differentiated Papillary Thyroid Carcinoma and in Patients With Thyroid Neoplasia of Unclear Malignant Potential
Brief Title: Sentinel Lymphnode in Patients With Papillary Thyroid Carcinoma and in Patients With Suspected Thyroid Neoplasia
Acronym: SNTC
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2009/71
Record Dates: First submitted 2010-03-16; First posted 2010-03-18 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Thyroid Neoplasms; Thyroid Cancer
Keywords: Sentinel node; Thyroid cancer; Thyroid neoplasia; Follicular neoplasia
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Papillary thyroid cancer: Patients with preoperatively diagnosed highly differentiated papillary thyroid cancer
  Interventions: Procedure: Histological investigation of the SN
- Tumour of uncertain malignant potential: Thyroid tumours with preoperative cytology indicating follicular neoplasia, or on cytology suspected but not proven malignancy
  Interventions: Procedure: Histological investigation of the SN

INTERVENTIONS:
Procedure: Histological investigation of the SN — 99m Tc- nanocolloid albumin, 10-15 MBq (volume 0.1-0.3 ml) is injected under ultrasound guidance in the thyroid tumour. Imaging (lymphoscintigraphy)with anterior and oblique projections is performed at 60 and 120 min after the injection. SN are mapped intraoperatively by a dedicated SN navigator and excised for final histology.

SUMMARY:
The standard surgical treatment for highly differentiated papillary thyroid cancer > 10 mm according to recent national and international guidelines, is total thyroidectomy and central lymphnode clearance, and for patients with cytology indicating thyroid neoplasia of unclear malignant potential hemithyroidectomy on the side of the tumour.

The study investigates if the sentinel lymphnode (SN)

* Reliably (with high sensitivity and specificity), can predict the pathological findings of the lymphnodes in the central compartment in patients with highly differentiated papillary thyroid cancer
* Is useful to aid in the final diagnosis and staging of thyroid neoplasias of unclear malignant potential, and could be used to select patients for further central lymphnode revision.

DETAILED DESCRIPTION:
The standard surgical treatment for highly differentiated papillary thyroid cancer > 10 mm according to recent national and international guidelines, is total thyroidectomy and central lymphnode clearance, and for patients with cytology indicating thyroid neoplasia of unclear malignant potential hemithyroidectomy on the side of the tumour.

There are however a number of clinical problems with these approaches:

* For patients with papillary thyroid cancer, a significant proportion will receive unnecessary extensive surgical treatment
* In papillary thyroid cancer, central lymphnode clearance increases the risk for complications, especially the risk for hypoparathyroidism.

According to a Scandinavian survey (Scandinavian Quality Register for Thyroid- and Parathyroid Surgery; www. thyroid-parathyroidsurgery.com),16 % of patients with unclear follicular neoplasia, will have a final histological diagnosis of thyroid cancer, and in half of them, this cancer will be of the papillary subtype. In patients with preoperatively suspected, but not proven malignancy by cytology, 30 % will receive a final histological diagnosis of thyroid cancer, and in these patients, 70 % will be of the papillary subtype. Typically these patients will undergo a second operation with a contralateral hemithyroidectomy. In many cases, due to risk for complications, central lymphnode clearance is avoided in these cases. Therefore, the staging of the cancer will be incomplete, and some patients will receive suboptimal surgical treatment.

The study is designed to compare SN investigation with the final histology of the central lymphnodes:

* Pretracheal and bilateral paratracheal for patients with preoperatively diagnosed papillary thyroid cancer
* Pretracheal and ipsilateral paratracheal for tumours of uncertain malignant potential on cytology

The identification of SN will be aided by preoperative ultrasound guided injection of 99m- Tc- nanocolloid albumin in the thyroid tumour. The results of the histological investigation of SN will be compared to that of the results from the central lymphnode clearance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with first time surgery for proven papillary thyroid cancer > 10 mm
* Patients with first time surgery for a cytologic diagnosis of follicular neoplasia or suspected (not proven) malignancy

Exclusion Criteria:

* Age below 18 years
* Pregnancy or lactation
* Inability to understand written and oral information or to comply with scheduled follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patients diagnosed and operated for papillary thyroid cancer > 10 mm at the Department of Surgery, Skåne University Hospital, Lund, Sweden
  _ Patients with diagnosed and operated for a thyroid tumour of unclear malignant potential at the Department of Surgery, Skåne University Hospital, Lund, Sweden
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-03; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of SN histology compared with the final histology of the non SN central lymph nodes (metastasis or no metastasis) | 14 days
  The histological investigation of the sentinel lymph node(s) (recorded as metastasis or no metastasis), will be compared to the definitive histological investigation of the non SN central lymphnodes (metastasis or no metastasis), cleared by surgery. Sensitivity and specificity of the histological SN investigation to predict the histological outcome of the non SN central lymphnodes (metastasis or no metastasis), will be calculated.

SECONDARY OUTCOMES:
Sensitivity of 99mTc-nanocolloid albumin in the diagnosis of a sentinel lymphnode | 1 day
  99mTc-nanocolloid albumin will be injected under guidence by ultrasonography. The sensitivity to detect a SN on preoperative imaging (detected SN on imaging/total number of investigations) and during surgery by a collimated probe for SN mapping(SN detected/total number of operations), will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Bergenfelz, MD, PhD, Principal Investigator — Department of Surgery, Skåne University Hospital, Lund
Locations (1):
- Department of Surgery and Department of Imaging, Skåne University Hospital, Lund, Sweden